CLINICAL TRIAL: NCT04197726
Title: Glycaemic Response to High REsistant STarch Bread
Acronym: REST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: QIB02/2019
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Blood Glucose Response
Keywords: Glycaemic response; Resistant starch; Bread

STUDY DESIGN:
Intervention Model Description: Double-blind randomised crossover study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sbeIIa/b white bread (Experimental): sbeIIa/b white bread with high resistant starch content
  Interventions: Other: sbeIIa/b white bread; Other: Control white bread
- Control white bread (Active Comparator): Reference white bread (wild-type)
  Interventions: Other: sbeIIa/b white bread; Other: Control white bread

INTERVENTIONS:
Other: sbeIIa/b white bread — one bread roll containing approximately 75 g of available carbohydrates to be consumed at breakfast
Other: Control white bread — one bread roll containing approximately 75 g of available carbohydrates to be consumed at breakfast

SUMMARY:
This study evaluates if the consumption of one sbeIIa/b white bread with high resistant starch content will result in a lower blood glucose response and increased satiety compared with reference white bread. All participants will be asked to consume once the sbeIIa/b white bread and the reference white bread during different visits.

DETAILED DESCRIPTION:
In an attempt to increase dietary fibre intake, research has focused on developing wheat-based food products with novel fibres and starches to complement fibre intake from whole grain foods. Resistant starch is starch that escapes digestion in the small intestine and may be fermented in the large intestine by the microbiota. Resistant starch is a type of dietary fibre and it is normally found in wheat-based foods made from refined flour but only in small amounts. White bread made from sbeIIa/b wheat, which has high levels of resistant starch (a type of fibre), is showing promise in modulating blood glucose response and increasing satiety compared with conventional white bread.

The primary aim of this study is to determine whether consumption of sbeIIa/b white bread at breakfast, gives rise to a lower postprandial blood glucose response compared with consumption of a reference white bread in healthy individuals.

Additional aims of the study include: determining whether consumption of sbeIIa/b white bread by healthy subjects, gives rise to a lower glucose concentration in interstitial fluid, as measured by a Continuous Glucose Monitoring system (CGM), compared with consumption of control white bread; and exploring satiety and energy intake changes in healthy individuals following consumption of sbeIIa/b white bread at breakfast, compared with consumption of control white bread.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Aged 18 to 65 years
* BMI between 18-25 kg/m2
* Non-smokers
* Those that live within a 40-mile radius of Norwich

Exclusion Criteria:

* Fasting glucose >6.1 mmol/L and/or HbA1c>42 mmol/mol, as assessed by a fasting blood test
* Eligibility screening results indicate they are not suitable to take part in this study
* Smokers (if they have smoked within the 6 weeks prior to the study or during the study)
* Suffer from allergy, intolerance, or sensitivity to gluten, yeast or any of the food ingredients used in this study
* Have a known allergy to adhesives that would prevent proper attachment of the Continuous Glucose Monitoring sensors
* Are pregnant and/or have been pregnant in the last year or are lactating and/or breastfeeding
* Are currently suffering from, or have ever suffered from eating disorders, any diagnosed gastrointestinal disease, gastrointestinal disorders including regular diarrhoea and constipation (excluding hiatus hernia unless symptomatic) or other inflammatory diseases like rheumatoid arthritis (RA), polymyalgia rheumatica or other connective tissues diseases
* Have undergone gastrointestinal surgery; this will be assessed on an individual basis
* Have been diagnosed with diabetes, anaemia as this may affect the study outcome
* Have been diagnosed with any long-term medical condition that may affect the study outcome (e.g. cardiovascular diseases, cancer)
* Regularly take over-the-counter medications for digestive/gastrointestinal conditions
* Use medications likely to interfere with energy metabolism, appetite regulation and hormonal balance, including long-term steroids, antibiotics. They may be able to participate if 4 weeks or more have passed from the end of a course such medication
* Regularly take laxatives (once a month or more) as this may affect blood glucose levels
* Take certain dietary supplements or herbal remedies and are unwilling to stop taking them (if required) for two weeks prior to and during the study period
* Are on, or plan to start, a diet programme that may affect the study outcome (e.g. 5:2 fasting diet) unless willing to abstain for 1 month prior to and during the study period
* Went through a weight change of ≥ 3kg in the preceding 2 months
* Have a recent history of substance abuse
* Regularly consume more than 14 units of alcohol a week
* Are unwilling to suspend smoking and vaping for the duration of the study.
* Are participating in another research project that involves dietary intervention or blood sampling.
* Are unwilling to provide GPs contact details
* Are related to or living with any member of the study team.
* Are unable to provide written informed consent
* Have not donated blood or taken part in another dietary intervention in the last 16 weeks and are unwilling to wait until 16 weeks have elapsed
* Those with abnormal blood pressure measurements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change in postprandial capillary glucose concentration | 3.5 hours
  Glucose concentration in capillary blood measured by finger prick test after the consumption of sbeIIa/b white bread compared to control white bread.
  Measurements will be taken during intervention visit 1 and 2 at -15, -10, -5, 15, 30, 45, 60, 75, 90, 120, 150, 180, 210 min.

SECONDARY OUTCOMES:
Change in postprandial glucose concentration in interstitial fluid | 4 hours
  Glucose concentration in interstitial fluid measured by continuous glucose monitoring system after the consumption of sbeIIa/b white bread compared to control white bread.
  Measurements will be taken during intervention visit 1 and 2 between -30 to 210 min.
Ad libitum intake | 2 hours
  Mean energy intake (kcal) at lunch after consumption of sbeIIa/b and control white bread.
  Measurements will be taken once during intervention visit 1 and 2.
Change in postprandial glucose concentration in interstitial fluid | 4 hours
  Glucose concentration in interstitial fluid measured by continuous glucose monitoring system after the consumption of ad libitum lunch to explore any second meal effects caused by prior intake of either sbeIIa/b white bread and control white bread at breakfast.
  Measurements will be taken during intervention visit 1 and 2 between 225 to 465 min.
Satiety | 3 hours
  Change of hunger feeling (appetite) will be examined using visual analog scale (0-10), 0 least and 10 greatest.
  Measurements will be taken during intervention visit 1 and 2, at 0, 32, 92, 182 min.
Sensory questionnaire | 30 minutes
  Sensory perception of sbeIIa/b white bread and control white bread will be evaluated using a nine-point hedonic scale to determine any differences overall acceptability based on specific attributes.
  A Just-About-Right (JAR) scale with five anchor points will be used to measure the appropriateness of the level of specific attributes to evaluate aroma, appearance, taste and texture of breads.
  Measurements will be taken once during intervention visit 1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Corrado, MSc, Principal Investigator — PhD student
Locations (1):
- Quadram Institute, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after publication in scientific journal within 18 months of study completion
Access Criteria: Data access will be reviewed by the study team